CLINICAL TRIAL: NCT06229353
Title: Developing and Evaluating a Novel Approach to Improve HPV Vaccination Coverage Among High-risk, Under-immunized Adults Via the Emergency Department
Status: Terminated | Type: Observational
Why Stopped: Slow pace of recruitment
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Andrzej Kulczycki, Associate Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300012035; MISP# 101971 (Other Grant/Funding Number: Merck Investigator Studies Program (MISP))
Record Dates: First submitted 2024-01-12; First posted 2024-01-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Human Papilloma Virus
Keywords: Gardasil 9; HPV
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine nonavalent; Papillomavirus Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Under-immunized Emergency Department adult patients: Adults attending the Emergency Department who are aged 18-45, without previous HPV vaccination history and without previously known infection from HPV high-risk strain, and in good functional capacity.
  Eligible participants will receive Gardasil 9 (HPV) vaccination if interested.
  Interventions: Biological: Gardasil 9

INTERVENTIONS:
Biological: Gardasil 9 — Prevent HPV-associated diseases and cancers
  Other Names: Human Papillomavirus Vaccine; HPV vaccine

SUMMARY:
To determine if the emergency department (ED) setting offers a viable space for improving HPV vaccination coverage among 18 to 45-year-old adults who have not yet received human papilloma virus (HPV) vaccination or who did not complete the vaccine series. This study will develop, pilot and evaluate an ED-based HPV vaccination protocol and program for ED patients aged 18-26 (for whom catch-up HPV vaccination is routinely recommended by the CDC) and separately for patients aged 27-45 (for whom it may be recommended under shared decision making, SDM).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years old
* in good functional capacity, as determined by the ED-attending clinician
* no known infection with HPV high risk strain types 6, 11, 16 and 18.

Exclusion Criteria:

* will not receive vaccine if participants lack mental clarity and if running a fever or in some pain.
* Patients aged <18 or > 45 years of age.
* Female patients with abnormal HPV results (including those with the high-risk HPV strain types 6, 11, 16, and 18) as determined by a previous PAP smear test or HPV test.
* Female patients who are known to be pregnant.
* Male patients with known cases of HPV-associated infections will also be excluded from the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pre-existing ED-patients in the waiting room who fit the eligibility criteria, as per the chart review which will indicate the participant's age, and if the participant is in good functional capacity, as determined by the ED-attending clinician, and if the participant has no known infection with HPV high risk strain types 6, 11, 16 and 18. Participants running fever or in pain at the time of the initial ED visit and still interested in receiving HPV vaccination, will be offered to come back for HPV vaccination when in good health at a later date.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Number of study participants who receive HPV vaccination at baseline | Baseline
  HPV vaccination will be administered at the time of the study participant's initial visit (baseline)
Number of study participants who receive HPV vaccination at 2 months | 2 months
  Number of study participants receiving dose 2 of the HPV vaccination series 2 months after initial study visit
Number of study participants who receive HPV vaccinations at 6 months | 6 months
  Number of study participants receiving dose 3 of the HPV vaccination series 6 months after initial study visit

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Kulczycki, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All Study data and results will be owned by the University of Alabama at Birmingham (UAB). UAB agrees that all Study data and results generated during the course of the Study may be used fully by Merck for any legitimate business purpose without any additional payments being made to UAB or the PI. Merck agrees not to publish the research data and results generated during the Study until the PI's publication or presentation of the Study results in accordance with Article 9, or 18 months following study completion or termination of this Agreement, whichever occurs first. Merck may disclose the research data and results to health authorities if such disclosure is prior to publication. Merck shall use reasonable efforts to disclose such research data and results confidentially. UAB agrees not to provide any commercial third party with access to or with the right to use the unpublished data or results for any purpose without Merck's permission which shall not be unreasonably withheld.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Article 9, or eighteen (18) months following completion of the Study or termination of this Agreement, whichever occurs first.